CLINICAL TRIAL: NCT03354871
Title: Developing Models for Fatigue Monitoring in Obstetrics and Gyne- Cology Residents Using Wearables
Acronym: IoT4Resident
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: International Business Machines (IBM) (Industry)
Responsible Party: Sponsor
Other Study IDs: 0081-17-HYMC
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is set out to observe heart-rate and related bio-metric indicators in Obstetrics and Gynecology residents during their duty hours, together with self-reporting of fatigue and tasks performances, in order to model possible relationships between the two.

DETAILED DESCRIPTION:
There are vast evidences of the harmful consequences of fatigue in medical residents, consequently, leading to poor task performances and in some cases may cause injury to the patients. Medically, fatigue is a non-specific symptom, which means that it has many possible causes and accompanies many different conditions. Elevated fatigue is an indication that a person may not be fit-to-task (i.e., task efficacy).The investigators main goal is to use readily available body-worn sensors, such as an activity wrist-band, to continuously monitor for fatigue as a possible antecedent to predictions of task-efficacy in the area of Obstetrics and Gynecology. This study is anchored in prior research which established basic models that correlate between heart-rate variability (HRV) and fatigue. Specific to this study, the investigators would like to further establish the validity of such models at the individual level, also with the perspective of fatigue as an early predictor of task performance related to practices in Obstetrics and Gynecology. The investigators aim is to extend HRV based models with additional personal measures (e.g., age, weight, activity level), possibly with the extraction of additional data-driven features, to improve model accuracy at the individual level. The investigators will also try to find relationships between such measurements and task effectiveness via the gathering of self-reports regarding on-the-job task performances.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be chosen from the obstetrics and gynecology department in the Hillel Yaffe medical center.

Exclusion Criteria:

* Chronic fatigue syndrome
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Obstetrics and gynecology residents in duty
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Fatigue determination model. | Through study completion, an average of 1 year.
  A model for detecting abnormal fatigue alert.

SECONDARY OUTCOMES:
Fatigue based fit-to-task model. | Through study completion, an average of 1 year.
  Model for estimation of for seen task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Hallak, M.D, Principal Investigator — Department of Obstetrics & Gynecology, Hillel Yaffe Medical Center, Hadera
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bundele, Mahesh M., and Rahul Banerjee.
- [Background] Szypulska, Małgorzata, and Zbigniew Piotrowski.